CLINICAL TRIAL: NCT02209571
Title: Exhaled Breath Analysis by Secondary Electrospray Ionisation Mass Spectrometry (SESI-MS) in Adults With Cystic Fibrosis: An Exploratory Matched Case-Control Study
Brief Title: Breath Analysis in in Adults With Cystic Fibrosis (CF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: KEK-ZH-Nr. 2014-0076
Record Dates: First submitted 2014-07-18; First posted 2014-08-06 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Cystic Fibrosis
Keywords: Breath Tests
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cystic Fibrosis (Experimental): Breath test and venous blood markers in cystic fibrosis patients
  Interventions: Other: Venous blood markers
- Control (Active Comparator): Breath test and venous blood markers in healthy subjects
  Interventions: Other: Venous blood markers

INTERVENTIONS:
Other: Venous blood markers — Routine venous blood sampling

SUMMARY:
Exploratory comparative evaluation of exhaled breath composition in cystic fibrosis patients with age and gender-matched healthy adults in order to identify a disease-specific exhaled breath pattern as well as to gain insight into pathophysiological and microbial contributions to exhaled breath composition.

DETAILED DESCRIPTION:
Although there is some evidence that breath composition reflects aspects of CF pathology, so far a disease-specific molecular breath profile has not been identified. Real-time, whole breath analysis incorporating all of the thousands of potentially relevant volatile compounds is needed in order to identify reliable CF-specific breath patterns. These may be used in future clinical applications to greatly enhance cost-effectiveness and simplicity of diagnostic testing for CF.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cystic fibrosis (for CF-patients)
* Age ≥ 18 years

Exclusion Criteria:

* Previous lung transplantation (for CF-patients)
* Pulmonary exacerbation within the preceding 6 weeks (for CF-patients)
* Moribund or severe disease prohibiting protocol adherence (for CF-patients)
* Respiratory illness requiring physician consultation within the preceding 6 weeks (for controls)
* Chronic respiratory illness (for controls)
* Physical or intellectual impairment precluding informed consent or protocol adherence
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Molecular composition of exhaled breath analysed by Secondary Electrospray Ionisation Mass Spectrometry (SESI-MS) | up to 2 years
  Breathprints (exhalome) molecular composition expressed in intensity patterns (so-called mass-to-charge or m/z pairs)

SECONDARY OUTCOMES:
Composite of clinical records | up to 2 years
  Clinical data assessed via questionaire, venous blood markers (clinical routine markers), sputum culture results (clinical routine bacteriology) (results to be reported as a single value for each Arm/Group)

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Kohler, MD, Prof, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Pulmonary Division, Zurich, Canton of Zurich, Switzerland